CLINICAL TRIAL: NCT03511612
Title: Comparison of the Ankle-Brachial Index Measurement Using a Specific Oscillometric Device vs. the Doppler Method
Acronym: ABIOSCILLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RC17_0075 (ABIOSCILLO)
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Arterial Disease, Ankle Brachial Index, Doppler
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pattern A (Other): Intervention : Each subject has 3 measurements of ABI starting with oscillometric device and then using the Doppler method.
  Interventions: Diagnostic Test: Measure ankle brachial index (ABI)
- Pattern B (Other): Intervention : Each subject has 3 measurements of ABI starting with Doppler method and then using oscillometric device.
  Interventions: Diagnostic Test: Measure ankle brachial index (ABI)

INTERVENTIONS:
Diagnostic Test: Measure ankle brachial index (ABI) — This is a head-to-head comparison of 2 methods of determination of the ABI, taking the Doppler method as the standard and the oscillometric device AVP as the challenger

SUMMARY:
Several methods are available to measure ankle brachial index (ABI) non-invasively. A recent scientific statement of the AHA considers the Doppler method as the reference. However because Doppler devices are not widely available in primary care, several attempts have been made to propose alternative methods, among whom oscillometric methods (automatic blood pressure machines) have attracted most attention.

We hypothesize that:

- the diagnostic characteristics (i.e. sensitivity, specificity and AUC) of the oscillometric method would be very good as compared to the Doppler method.

the oscillometric method would have better intra- and inter-observer reproducibilities as compared to the Doppler method.

ELIGIBILITY:
Inclusion Criteria:

Patients referred with the suspicion of PAD, either because of:

* symptoms in favor of intermittent claudication or more atypical pain when walking, or
* asymptomatic individuals with the presence of at least 2 cardiovascular risk factors among the following :

  * Men > 60 years or women > 65 years
  * Regular cigarette smoking >10 years, either current or in the past
  * Treated Type-2 diabetes >5 years or Type-1 diabetes >20 years
  * Treated hypertension
  * High blood cholesterol (either total-C >240 mg/dl or LDL-C >160 mg/dl) or treated by statins or other lipid-lowering agents
  * Documented history of coronary artery disease (history of PCI or CABG, or previous myocardial infarction, or CAD documented by coronary angiography)
  * Documented history of ischemic stroke

Exclusion Criteria:

* Patients with revascularized PAD
* Patients with critical limb ischemia or leg/foot ulcers
* Cardiac arrhythmia: Atrial fibrillation, atrial flutter, frequent supra- and ventricular ectopic beats
* Patients under dialysis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Measurement of the ABI | Day of the inclusion
  Measurement of the ABI, with Doppler method as reference

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, France

REFERENCES:
- [Background] Ichihashi S, Desormais I, Hashimoto T, Magne J, Kichikawa K, Aboyans V. Accuracy and Reliability of the Ankle Brachial Index Measurement Using a Multicuff Oscillometric Device Versus the Doppler Method. Eur J Vasc Endovasc Surg. 2020 Sep;60(3):462-468. doi: 10.1016/j.ejvs.2020.06.013. Epub 2020 Aug 3. PMID 32763120